CLINICAL TRIAL: NCT01485315
Title: Effects of Red Blood Cell Transfusion on Mortality and Morbidity in Patients With Septic Shock
Brief Title: Transfusion-requirements in Septic Shock Trial
Acronym: TRISS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scandinavian Critical Care Trials Group (Other)
Collaborators: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Rigshospitalet, Denmark (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Anders Perner, Principle Investigator, Scandinavian Critical Care Trials Group
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-3-2011-114
Record Dates: First submitted 2011-11-30; First posted 2011-12-05 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Blood Transfusion; Erythrocyte Count

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liberal blood transfusion (Active Comparator): Blood transfusion at haemoglobin 9.0 g/dl (5.6 mM) or less
  Interventions: Biological: SAGM (Saline-Adenine-Glucose-Mannitol) blood transfusion
- Restrictive blood transfusion (Active Comparator): Blood transfusion at haemoglobin 7.0 g/dl (4.3 mM) or less
  Interventions: Biological: SAGM (Saline-Adenine-Glucose-Mannitol) blood transfusion

INTERVENTIONS:
Biological: SAGM (Saline-Adenine-Glucose-Mannitol) blood transfusion — One unit prestorage, leuko-depleted SAGM blood at haemoglobin at 9.0 g/dl (5.6 mM) or less at point-of-care testing
  Other Names: Liberal red blood cell (RBC) transfusion
  Arms: Liberal blood transfusion
Biological: SAGM (Saline-Adenine-Glucose-Mannitol) blood transfusion — One unit prestorage, leuko-depleted SAGM blood at haemoglobin 7.0 g/dl (4.3 mM) or less at point-of-care testing
  Other Names: Restrictive red blood cell (RBC) transfusion
  Arms: Restrictive blood transfusion

SUMMARY:
Patients with blood poisoning - sepsis - often receive blood transfusions in the intensive care unit. The evidence that blood transfusion leads to improved outcome is limited and the blood may be harmful to some of these patients. To bridge the gap between clinical practice and evidence, a large randomised clinical trial is needed to document the efficacy and safety of RBC transfusion in these very sick patients

DETAILED DESCRIPTION:
Background Septic patients often receive red blood cell (RBC) transfusions in the intensive care unit. The evidence that RBC transfusion leads to improved outcome is limited and the intervention may be harmful to some of these patients. In contrast, current guidelines recommend restrictive transfusion of RBC for critical ill patients without septic shock. To bridge the gap between clinical practice and evidence, a large randomised clinical trial is needed to document the efficacy and safety of RBC transfusion in patients with septic shock

Design Pragmatic, multicenter, randomised, outcome assessment-blinded trial of patients with septic shock to RBC transfusion at haemoglobin (Hb) transfusion trigger of 7 g/dl (4.4 mM) or 9 g/dl (5.6 mM), stratified by the presence of haematological malignancy and centre.

Inclusion and exclusion criteria:

To increase the validity of the trial inclusion criteria will be broad with few exclusions

Outcome measures The outcome measures will mainly be patient-important but ICU- and hospital length of stay will also be assessed

Trial size 2 x 500 patients will be needed to show a 9% absolute risk difference in 90-day mortality (baseline mortality of 45%, relative risk reduction 20% (from septic patients in the TRICC trial), alpha of 0.05 (two-sided) and a beta of 0.20 that is a power of 80% (1-beta).

An interim-analysis will be performed after 500 patients. The Data Safety and Monitoring Board (DMSC) will recommend that the trial is stopped if a group-difference in 90-day mortality with p<0.001.

Time Line The first patient is expected to be randomised December 1st 2011 and the trial database is expected to be closed early 2014. The main manuscript will be submitted shortly thereafter.

Funding The trial is publicly funded by the Danish Strategic Research Council

ELIGIBILITY:
Inclusion Criteria:

* Patient in the ICU AND
* Fulfil the criteria for septic shock AND
* Have haemoglobin of 9.0 g/dl (5.6 mM) or less AND
* Consent obtainable from patient or proxy or national law allows delayed consent

Exclusion Criteria:

* Documented wish against transfusion OR
* Previous serious adverse reaction with blood product OR
* Acute coronary syndrome OR
* Life-threatening bleeding OR
* RBC transfusion during current ICU admission OR
* Withdrawal from active therapy or brain death OR
* Lack of informed consent (depending on national law) OR
* Acute burn injury regardless of degree and burn surface area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1005 (Actual)
Dates: Start 2011-11; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Mortality | 90 day
  All cause 90 day mortality

SECONDARY OUTCOMES:
Persistent organ failure | Day 5
  Defined as need for ventilation, vasopressor/inotrope infusion or renal replacement therapy
Persistent organ failure | Day 14
  Defined as need for ventilation, vasopressor/inotrope infusion or renal replacement therapy
Persistent organ failure | Day 28
  Defined as need for ventilation, vasopressor/inotrope infusion or renal replacement therapy
Anaphylactic/allergic reactions | Followed up until ICU discharge; an expected average of one week
  Defined by the clinician on the basis of mucocutaneous signs and symptoms (e.g. urticaria, pruritus, localised angio- oedema).
Haemolytic complications after transfusion of RBC | Followed up until ICU discharge; an expected average of one week
  Defined by the clinician on the basis of haemoglobinuria or increased free plasma haemoglobin.
Transfusion associated acute lung injury (TRALI) | Followed up until ICU discharge; an expected average of one week
  TRALI defined as:
  I. Acute or worsening hypoxaemia ((PaO2/FiO2 < 40 (PaO2 in kPa) or <300 (PaO2 in mmHg) regardless of PEEP) OR > 50% relative increase in FiO2.
  AND II. Occurrence within 6 hours after RBC transfusion AND III. Acute or worsening pulmonary infiltrates on frontal chest x-ray OR clinical signs of overt pulmonary oedema
Transfusion associated circulatory overload (TACO) | Followed up until ICU discharge; an expected average of one week
  TACO defined as:
  I. Acute or worsening hypoxaemia ((PaO2/FiO2 < 40 (PaO2 in kPa) or <300 (PaO2 in mmHg) regardless of PEEP) OR > 50% relative increase in FiO2.
  AND II. Occurrence within 6 hours after RBC transfusion AND III. Acute or worsening pulmonary infiltrates on frontal chest x-ray OR clinical signs of overt pulmonary oedema AND IV. Increased blood pressure AND VI. Positive fluid balance
Ischaemic events | Followed up until ICU discharge; an expected average of one week
  Defined as either myocardial, cerebral, intestinal or acute limb ischaemia
Days alive without life support | 90-days
  Life support defined as need for ventilation, vasopressor/inotrope infusion or renal replacement therapy. Days alive without each of these interventions will be reported
Days alive and out of hospital | 90 days
Mortality within the whole observation period | One year after randomisation of the last patient
  Mortality within the whole observation period reported at day 28, six-month and 1 year after randomisation of the last patient.
Health-related quality of life | 1 year
  Physical and mental component summary scores of SF 36

CONTACTS AND LOCATIONS:
Overall Officials: Anders Perner, MD, PhD, Principal Investigator — Dept. of Intensive Care, Rigshospitalet / SCCTG
Locations (32):
- Denmark (19):
  - Ålborg University Hospital, Aalborg
  - Aarhus University Hospital, NBG, Aarhus
  - Aarhus University Hospital, Skejby, Aarhus
  - Bispebjerg Hospital, Copenhagen
  - Glostrup Hospital, Copenhagen
  - Hvidovre Hospital, Copenhagen
  - Rigshospitalet, Copenhagen
  - Gentofte Hospital, Gentofte Municipality
  - Herning Hospital, Herning
  - Hjørring Hospital, Hjørring
  - Holbæk Hospital, Holbæk
  - Horsens Hospital, Horsens
  - Kolding Hospital, Kolding
  - Køge Hospital, Køge
  - Næstved Hospital, Næstved
  - Randers Hospital, Randers
  - Slagelse Hospital, Slagelse
  - Sønderborg Hospital, Sønderborg
  - Vejle Hospital, Vejle
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Joensuu Hospital, Joensuu
  - Tampere University Hospital, Tampere
- Norway (4):
  - Ålesund Hospital, Ålesund
  - Haukeland University Hospital, Bergen
  - Akershus University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
- Sweden (6):
  - Halmstad Hospital, Halmstad
  - Helsingborg Hospital, Helsingborg
  - Karolinska Hospital, Huddinge, Stockholm
  - Karolinska Institutet Solna, Stockholm
  - Södersjukhuset, Stockholm
  - Växjö Hospital, Vaxjo

REFERENCES:
- [Background] Holst LB, Haase N, Wetterslev J, Wernerman J, Aneman A, Guttormsen AB, Johansson PI, Karlsson S, Klemenzson G, Winding R, Nebrich L, Albeck C, Vang ML, Bulow HH, Elkjaer JM, Nielsen JS, Kirkegaard P, Nibro H, Lindhardt A, Strange D, Thormar K, Poulsen LM, Berezowicz P, Badstolokken PM, Strand K, Cronhjort M, Haunstrup E, Rian O, Oldner A, Bendtsen A, Iversen S, Langva JA, Johansen RB, Nielsen N, Pettila V, Reinikainen M, Keld D, Leivdal S, Breider JM, Tjader I, Reiter N, Gottrup U, White J, Wiis J, Andersen LH, Steensen M, Perner A. Transfusion requirements in septic shock (TRISS) trial - comparing the effects and safety of liberal versus restrictive red blood cell transfusion in septic shock patients in the ICU: protocol for a randomised controlled trial. Trials. 2013 May 23;14:150. doi: 10.1186/1745-6215-14-150. PMID 23702006
- [Result] Holst LB, Haase N, Wetterslev J, Wernerman J, Guttormsen AB, Karlsson S, Johansson PI, Aneman A, Vang ML, Winding R, Nebrich L, Nibro HL, Rasmussen BS, Lauridsen JR, Nielsen JS, Oldner A, Pettila V, Cronhjort MB, Andersen LH, Pedersen UG, Reiter N, Wiis J, White JO, Russell L, Thornberg KJ, Hjortrup PB, Muller RG, Moller MH, Steensen M, Tjader I, Kilsand K, Odeberg-Wernerman S, Sjobo B, Bundgaard H, Thyo MA, Lodahl D, Maerkedahl R, Albeck C, Illum D, Kruse M, Winkel P, Perner A; TRISS Trial Group; Scandinavian Critical Care Trials Group. Lower versus higher hemoglobin threshold for transfusion in septic shock. N Engl J Med. 2014 Oct 9;371(15):1381-91. doi: 10.1056/NEJMoa1406617. Epub 2014 Oct 1. PMID 25270275
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836